CLINICAL TRIAL: NCT00619294
Title: Digital Tonometry for Measurement of Peripheral Artery Reactive Hyperemia as Non-invasive Test for Diagnosis of Coronary Artery Spasm
Brief Title: Endothelial Dysfunction and Coronary Artery Spasm
Status: Completed | Type: Observational
Sponsor: Kumamoto University (Other)
Responsible Party: Principal Investigator, Seigo Sugiyama, MD, PhD, Kumamoto University
Other Study IDs: 743
Record Dates: First submitted 2008-02-08; First posted 2008-02-20 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-09

CONDITIONS: Coronary Vasospasm
Keywords: Coronary Vasospasm; Endothelium, Vascular; Vasodilation; Hyperemia
MeSH Terms: conditions — Coronary Vasospasm; Aneurysm; Hyperemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Non-obstructive coronary artery disease (NOCAD) frequently accounts for myocardial ischemia in women. Endothelial dysfunction is a pathogenic factor in coronary spastic angina (CSA). CSA is an important cause of NOCAD diagnosed invasively by coronary angiography (CAG). Digital reactive hyperemia peripheral arterial tonometry (RH-PAT) provides noninvasive evaluation of endothelial dysfunction. The investigators hypothesized that the fingertip RH-PAT could predict the presence of CSA in women.

DETAILED DESCRIPTION:
Outline of methods:

RH-PAT was measured in women with chest pain prior to CAG. Coronary spasm was diagnosed by intra-coronary acetylcholine (ACh) provocation test. Using Flow-Wire, we assessed coronary endothelial function by coronary blood flow increase in response to ACh (ACh-CBF) and coronary flow reserve was assessed by adenosine (Ad-CFR).

ELIGIBILITY:
Inclusion Criteria:

* Stable post-menopausal women complaining angina-like chest pain

Exclusion Criteria:

* Severe valvular disease
* Hypertrophic cardiomyopathy
* Severe peripheral artery disease
* Uncontrolled hypertension
* Severe collagen diseases
* Acute coronary syndrome

Ages: 40 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kumamoto University Hospital
Sampling Method: Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2006-08; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Ischemic heart disease diagnosed by cardiac catheterization | From Aug 2006 to May 2009

CONTACTS AND LOCATIONS:
Locations (1):
- Kumamoto University Hospital, Kumamoto, Kumamoto, Japan

REFERENCES:
- [Derived] Matsuzawa Y, Sugiyama S, Sugamura K, Nozaki T, Ohba K, Konishi M, Matsubara J, Sumida H, Kaikita K, Kojima S, Nagayoshi Y, Yamamuro M, Izumiya Y, Iwashita S, Matsui K, Jinnouchi H, Kimura K, Umemura S, Ogawa H. Digital assessment of endothelial function and ischemic heart disease in women. J Am Coll Cardiol. 2010 Apr 20;55(16):1688-96. doi: 10.1016/j.jacc.2009.10.073. PMID 20394872